CLINICAL TRIAL: NCT05563779
Title: Mode Of Ventilation During Critical Illness Pilot Trial
Acronym: MODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kevin P Seitz, Clinical Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 220446
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: In the MODE trial, the entire study ICU will be assigned to a single mode for continuous mandatory ventilation and the ICU will switch between volume control, pressure control, and adaptive pressure control every month in a randomly generated sequence (cluster-crossover).
Who Masked: Outcomes Assessor
Masking Description: Observer bias will be minimized by use of objective endpoints collected in duplicate by [1] study personnel blinded to group assignment and [2] automated data extraction from the electronic health record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volume Control mode (Active Comparator): During invasive mechanical ventilation in a study location, Volume Control will be used as the mode for continuous mandatory ventilation.
  Interventions: Other: Volume Control mode
- Pressure Control mode (Active Comparator): During invasive mechanical ventilation in a study location, Pressure Control will be used as the mode for continuous mandatory ventilation.
  Interventions: Other: Pressure Control mode
- Adaptive Pressure Control mode (Active Comparator): During invasive mechanical ventilation in a study location, Adaptive Pressure Control will be used as the mode for continuous mandatory ventilation.
  Interventions: Other: Adaptive Pressure Control mode

INTERVENTIONS:
Other: Volume Control mode — Volume Control mode for mechanical ventilation
  Arms: Volume Control mode
Other: Pressure Control mode — Pressure Control mode for mechanical ventilation
  Arms: Pressure Control mode
Other: Adaptive Pressure Control mode — Adaptive Pressure Control mode for mechanical ventilation
  Arms: Adaptive Pressure Control mode

SUMMARY:
Landmark trials in critical care have demonstrated that, among critically ill adults receiving invasive mechanical ventilation, the use of low tidal volumes and low airway pressures prevents lung injury and improves patient outcomes. Limited evidence, however, informs the best method of mechanical ventilation to achieve these targets. To provide mechanical ventilation, clinicians must choose between modes of ventilation that directly control tidal volumes ("volume control"), modes that directly control the inspiratory airway pressure ("pressure control"), and modes that are hybrids ("adaptive pressure control"). Whether the choice of the mode used to target low tidal volumes and low inspiratory plateau pressures affects clinical outcomes for critically ill adults receiving mechanical ventilation is unknown. All three modes of mechanical ventilation are commonly used in clinical practice. A large, multicenter randomized trial comparing available modes of mechanical ventilation is needed to understand the effect of each mode on clinical outcomes. The investigators propose a 9-month cluster-randomized cluster-crossover pilot trial evaluating the feasibility of comparing three modes (volume control, pressure control, and adaptive pressure control) for mechanically ventilated ICU patients with regard to the outcome of days alive and free of invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Receiving mechanical ventilation through an endotracheal tube or tracheostomy
* Admitted to the study ICU

Exclusion Criteria:

* Patient is pregnant
* Patient is a prisoner
* Patient receiving invasive mechanical ventilation at place of residence prior to hospital admission
* Patient receiving extracorporeal membrane oxygenation at the time of admission to the study ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days (VFDs) to day 28 after enrollment | Enrollment to 28 days
  Number of days alive and free from invasive mechanical ventilation between the final liberation from invasive mechanical ventilation before 28 days and study day 28. Patients who continue to receive invasive mechanical ventilation at day 28 or have died prior to day 28 will receive zero VFDs. For patients who return to invasive mechanical ventilation and are subsequently liberated from invasive mechanical ventilation prior to day 28, VFDs will be counted from final liberation from mechanical ventilation.

OTHER OUTCOMES:
Exposure to assigned study mode in first 3 days (Feasibility Outcome) | Enrollment to 72 hours
  Proportion of time in the assigned mode while receiving invasive mechanical ventilation in the study ICU between enrollment and 72 hours after enrollment
Adherence to study mode in first 3 days (Feasibility Outcome) | Enrollment to 72 hours
  Proportion of time in the assigned mode while receiving invasive mechanical ventilation in the study ICU with a mandatory mode between enrollment and 72 hours after enrollment (excluding time spent in spontaneous modes)
Time from enrollment to initiation of assigned mode of mechanical ventilation (Feasibility Outcome) | Enrollment to 28 days
Number of patients with a "Mode Modification Sheet" completed by treating clinicians (Feasibility Outcome) | Enrollment to 28 days
Median daily exhaled tidal volume (mL/kg predicted body weight) on each study day (Exploratory Efficacy and Safety Outcome) | Enrollment to 7 days
Exhaled tidal volumes above target range (Exploratory Efficacy and Safety Outcome) | Enrollment to 7 days
  Proportion of recorded breaths with exhaled tidal volume values above target range (>8mL/kg predicted body weight) on each study day
Hypoxemia during mechanical ventilation (Exploratory Safety and Efficacy Outcome) | Enrollment to 28 days
  Episodes of hypoxemia during mechanical ventilation: SpO2 <85% for more than 5 minutes
Severe acidemia during mechanical ventilation (Exploratory Safety and Efficacy Outcome) | Enrollment to 28 days
  Episodes of severe acidemia during mechanical ventilation: pH < 7.1 on blood gas
Number of blood gas laboratory tests per day while receiving mechanical ventilation (Exploratory Safety and Efficacy Outcome) | Enrollment to 28 days
Pneumomediastinum or pneumothorax during course of mechanical ventilation (Exploratory Efficacy and Safety Outcome) | Enrollment to 28 days
SOFA score daily on the first 7 study days (Exploratory Safety and Efficacy Outcome) | Enrollment to 7 days
Delirium and coma free days to day 28 (Exploratory Efficacy and Safety Outcome) | Enrollment to 28 days
  Number of days alive and without delirium or coma before 28 days to study day 28
Intensive care unit-free days to study day 28 (Exploratory Clinical Outcome) | Enrollment to 28 days
  Number of days alive and free from intensive care unit admission after the final transfer out of the intensive care unit before 28 days to study day 28
Hospital-Free days to study day 28 (Exploratory Clinical Outcome) | Enrollment to 28 days
  Number of days alive and free from hospitalization after the final transfer out of the hospital before 28 days to study day 28
In-hospital mortality to study day 28 (Exploratory Clinical Outcome) | Enrollment to 28 days
  All-cause mortality prior to discharge from the hospital, assessed at 28 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P. Seitz, MD, MSc, Principal Investigator — Clinical Fellow
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of primary trial results and will remain available for at least 5 years.
Access Criteria: Following publication, individual patient data will be made available for sharing to researchers with 1) a signed data access agreement, 2) research testing a hypothesis, 3) a protocol that has been approved by an institutional review board, and 4) a proposal that has received approval from the principal investigator.
  Even though the final dataset will be stripped of identifiers prior to release for sharing, the inherent link between the period in which the patient was admitted to the study ICU and group assignment in a cluster-crossover trial introduces a significant risk for deductive disclosure of subjects. Thus, we will make the data available to users only under a data sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Seitz KP, Lloyd BD, Wang L, Shotwell MS, Qian ET, Muhs AL, Richardson RK, Rooks JC, Hennings-Williams V, Sandoval CE, Richardson WD, Morgan TL, Thompson AN, Hastings PG, Ring TP, Stollings JL, Talbot EM, Krasinski DJ, DeCoursey BR, Marvi TK, DeMasi SC, Gibbs KW, Self WH, Mixon AS, Rice TW, Semler MW, Casey JD; Pragmatic Critical Care Research Group. Effect of Ventilator Mode on Ventilator-Free Days in Critically Ill Adults: A Randomized Clinical Trial. Chest. 2025 Oct;168(4):912-923. doi: 10.1016/j.chest.2025.03.024. Epub 2025 Apr 4. PMID 40189043
- [Derived] Seitz KP, Lloyd BD, Wang L, Shotwell MS, Qian ET, Richardson RK, Rooks JC, Hennings-Williams V, Sandoval CE, Richardson WD, Morgan T, Thompson AN, Hastings PG, Ring TP, Stollings JL, Talbot EM, Krasinski DJ, Decoursey B, Gibbs KW, Self WH, Mixon AS, Rice TW, Semler MW, Casey JD. Protocol and Statistical Analysis Plan for the Mode of Ventilation During Critical Illness (MODE) Trial. CHEST Crit Care. 2024 Mar;2(1):100033. doi: 10.1016/j.chstcc.2023.100033. Epub 2023 Nov 25. PMID 38742219
- [Derived] Seitz KP, Lloyd BD, Wang L, Shotwell MS, Qian ET, Richardson RK, Rooks JC, Hennings-Williams V, Sandoval CE, Richardson WD, Morgan T, Thompson AN, Hastings PG, Ring TP, Stollings JL, Talbot EM, Krasinski DJ, Decoursey B, Gibbs KW, Self WH, Mixon AS, Rice TW, Semler MW, Casey JD. Protocol and statistical analysis plan for the Mode of Ventilation During Critical IllnEss (MODE) trial. medRxiv [Preprint]. 2023 Jul 24:2023.07.21.23292998. doi: 10.1101/2023.07.21.23292998. PMID 37546787